CLINICAL TRIAL: NCT06448507
Title: Effectiveness of a Needle-free Local Anesthetic Technique Compared to the Traditional Syringe Technique for the Restoration of Primary Molars and Young Permanent Molars: A Single-blind Randomized Clinical Trial
Brief Title: Comparison of a Needle-free Local Anesthetic Technique With Traditional Syringe [ Needle Syringe] Technique for the Restoration of Primary Molars and Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, satish vishwanathaiah, Associate professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jazan University
Record Dates: First submitted 2024-05-17; First posted 2024-06-07 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Child Behaviour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INJEX (Experimental): needle less device
  Interventions: Device: INJEX [Needle less anesthesia]
- Needle syringe (Active Comparator): traditional dental needle
  Interventions: Device: Syringe Needle [ Traditional technique]

INTERVENTIONS:
Device: INJEX [Needle less anesthesia] — already described
  Arms: INJEX
Device: Syringe Needle [ Traditional technique] — described
  Arms: Needle syringe

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of needle free system and dental needle system [Traditional syringe system] for restoration of Primary and young permanent teeth. The main questions it aims to answer are:

1. To evaluate pain perception for restoration of primary and young permanent tooth with a needle free system in a pediatric population.
2. To evaluate pain perception for restoration of primary and young permanent tooth with needle syringe [Traditional syringe system] method in a pediatric population
3. Time required to deliver anesthesia using needle free system vs Needle syringe [ traditional syringe system]

Participants who enrolled in the study will be anesthetized according to the respective groups i,e needle free system and traditional dental needle system and restoration will be done.

DETAILED DESCRIPTION:
Before the start of the study a written informed consent and ascent was obtained from each parent of the children included in the study stating they accepted the treatment. Ethical clearance will be obtained before the start of the study. Patients reporting to the dental clinics, college of dentistry will be included in the study.

Sample size estimation:

the sample size was estimated to be twenty-one (21). Twenty percent of the estimated sample size was added to compensate for sampling loss if any, thus the final sample size accounted to a total of twenty-five (25) participants in each group.

study design: It was a single blinded randomized controlled trial

Randomization:

Children will be allocated into one of the following two groups using a simple randomization method with a random number table, employing the sequentially numbered opaque sealed envelopes method of allocation concealment.

Group I: All participants in this group were subjected to the traditional needle syringe system. Local infiltration of Scandicaine 2% Speciale [Mepivacaine Hydrochloride and adrenaline] was administered using a traditional needle syringe equipped with a 27-gauge needle.

Group II: Participants in this group received the needle-free injection system, specifically the INJEX (Injex Pharma AG, Germany) 0.3ml of 2% Scandicaine will be adminsitered.

Intervention procedure

To avoid any operator-related bias, a single operator will manage the entire anesthesia protocol for all participants in the trial. Employing the "tell-show-do" technique, all relevant treatment equipment and protocols were introduced and explained to the participants. The injection process was fully described using appropriate euphemisms. Before administering the injection, the treatment area at the injection site was cleansed using a sterile dry gauze, and a small amount of topical anesthetic (Benzocaine 20%, NJ, USA) was applied, remaining in place for at least one minute. Following the application of topical anesthesia, local anesthesia was administered based on the participant's assigned group. After a standard waiting period of three minutes for the onset of anesthesia, dental caries was removed, dycal applied and final restoration with composite was done.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 - 14 years
* Existence of deep carious Primary and Permanent molar, indicated for Indirect pup capping.
* Complete physical and mental health without any confounding medical history
* Parents who gave written informed consent

Exclusion Criteria:

* Children below 7 years of age
* Children complaining of irreversible pulpitis.
* Children with Negative behaviour according to the wright's modification of Frankl
* Behaviour Rating scale (FBRS) during initial examination
* Children with medical or mentally compromised

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Comfort and Patient acceptance of the needle less anesthesia technique and traditional/ syringe needle in children | during and immediately after the delivery of anesthesia
  FLACC assessment. FLACC gives an observational pain scale during the delivery of anesthesia
Comfort and Patient acceptance of the needle less anesthesia technique and traditional/needle syringe in children | During and immediately after the delivery of anesthesia
  Wong Baker Scale. Used to self-assess and effectively communicate the severity of pain they may be experiencing

SECONDARY OUTCOMES:
Comfort and Patient acceptance of the needle less anesthesia technique and traditional/needle syringe in children | before the delivery of anesthesia, during the delivery of anesthesia and after the delivery of anesthesia
  FBRS
Comfort and Patient acceptance of the needle less anesthesia technique and traditional/needle syringe in children | Before the delivery of anesthesia, immediately after the delivery of anesthesia, and 1 minute after the delivery of anesthesia
  Pulse rate
Comfort and Patient acceptance of the needle less anesthesia technique and traditional/needle syringe in children | during the delivery of anesthesia
  time of local anesthesia administration

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No